CLINICAL TRIAL: NCT00886132
Title: A Phase 2 Study of Sunitinib in Recurrent and/or Metastatic Adenoid Cystic Carcinoma of the Salivary Glands
Brief Title: A Study of Sunitinib in Recurrent and/or Metastatic Adenoid Cystic Carcinoma of the Salivary Glands
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACC-Siu 2006
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Adenoid Cystic Carcinoma; Salivary Gland Cancer
Keywords: Phase 2 Study; Sunitinib; Recurrent; Metastatic; Adenoid Cystic Carcinoma; Salivary Glands; Metastasis
MeSH Terms: conditions — Carcinoma, Adenoid Cystic; Salivary Gland Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib (Experimental): Patients with progressive, recurrent and/or metastatic ACC treated with sunitinib 37.5 mg daily in this single-arm, two-stage phase II trial.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — 37.5 mg taken orally, daily every 28-day cycles
  Other Names: Sutent, SU11248

SUMMARY:
This is a phase II study to evaluate the effectiveness of study drug sunitinib malate in patients with recurrent and/or metastatic adenoid cystic carcinomas of the salivary gland. There currently is not standard of care for this type of cancer and it has hoped that sunitinib will have antitumor effects on patients with this type of cancer.

DETAILED DESCRIPTION:
This is an open-label phase II study of sunitinib malate in patients with recurrent and/or metastatic adenoid cystic carcinomas (ACC) of major or minor salivary gland origin. Sunitinib is a novel, multi-targeted small molecule inhibitor of the receptor tyrosine kinases (RTKs), including vascular endothelial growth factor receptors (VEGFs), platelet derived growth factor receptors (PDGFRs) and stem cell factor receptor (KIT), that are involved in tumour proliferation and angiogenesis. VEGF expression has been associated clinically with disease prognosis in many different types of cancers and a number of studies have suggested that VEGF may play an important role in the pathogenicity of ACC. Sunitinib is expected to inhibit PDGF- and VEGF-driven angiogenesis and, as a consequence, limit solid tumour growth.This study will determine the anti-tumour activity of sunitinib in ACC of the salivary glands using objective response rates (partial and complete responses) as its primary objective.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic or cytologic adenoid cystic carcinomas of major or minor salivary gland origin.
* Patients must have recurrent and/or metastatic disease that is progressive and not amenable to surgery or curative radiotherapy occurring within 6 months of study entry:

  * at least a 20% increase in radiologically or clinically measurable disease;
  * appearance of any new lesions or
  * deterioration in clinical status
* Patients must have measurable disease, at least one lesion that can be accurately measured in at least one dimension as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
* Patients with prior therapy with at least a 4 weeks' interval between any chemotherapy (6 weeks for nitrosoureas or mitomycin C), radiotherapy or surgery and study enrollment. Exceptions may be made for low dose, non-myelosuppressive radiotherapy.
* Patients must be 18 years of age or older.
* Life expectancy of greater than 12 weeks.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes >3,000/μL
  * absolute neutrophil count >1,500/μL
  * platelets >100,000/μL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤2.5 X institutional upper limit of normal
  * amylase/lipase within normal institutional limits
  * creatinine within normal institutional limits
  * creatinine clearance >60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Cardiac ejection fraction within the institutional range of normal as measured by ECHO or MUGA scan.
* Patients must have QTc < 500 msec on baseline ECG.
* Patients with New York Heart Association (NYHA) Class II cardiac function:

  * with a history of Class II heart failure who are asymptomatic on treatment
  * with prior anthracycline exposure
  * who have received central thoracic radiation that included the heart in the radiotherapy port.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier. At least 4 weeks must have elapsed since any major surgery.
* Patients receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib.
* Patients with QTc prolongation or other significant ECG abnormalities.
* Patients with poorly controlled hypertension.
* Patients who require use of therapeutic doses of coumarin-derivative anticoagulants such as warfarin, although doses of up to 2 mg daily are permitted for prophylaxis of thrombosis. Note: Low molecular weight heparin is permitted provided the patient's PT INR is <1.5.
* Patients with any condition that impairs their ability to swallow and retain sunitinib tablets.
* Patients with any of the following conditions:

  * Serious or non-healing wound, ulcer, or bone fracture.
  * History of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess within 28 days of treatment.
  * Any history of cerebrovascular accident or transient ischemic attack within 12 months prior to study entry.
  * History of myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within 12 months prior to study entry.
  * History of pulmonary embolism within the past 12 months.
  * Class III or IV heart failure as defined by the NYHA.
* Patients taking medications that are potent inducers or inhibitors of the CYP3A4 liver enzyme (unless deemed acceptable by the Principal Investigator).
* Patients with a pre-existing thyroid abnormality who are unable to maintain thyroid function in the normal range with medication.
* Patients with known brain metastases.
* Patients with uncontrolled intercurrent illness including, ongoing or active infections or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women. Breastfeeding should be discontinued if the mother is treated with sunitinib.
* HIV-positive patients on combination antiretroviral therapy
* Patients taking any of the medications that may cause QTc prolongation unless the required washout period has been met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To determine the antitumor activity of sunitinib in recurrent and/or metastatic adenoid cystic carcinoma of the salivary glands using objective response rates (partial and complete responses). | Changes in tumor measurements must be confirmed by repeat assessments that should be performed not less than 4 weeks after the criteria for response are first met.

SECONDARY OUTCOMES:
To determine the duration of objective response, rate and duration of stable disease, progression-free, median and overall survival rates of sunitinib in recurrent and/or metastatic adenoid cystic carcinoma of the salivary glands. | From the time measurement criteria are met for CR or PR until the first date that recurrent or progressive disease is objectively.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Hotte, MD, Principal Investigator — Juravinski Cancer Centre
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada